CLINICAL TRIAL: NCT05573165
Title: A Pilot Study of the Effects of 4 vs 3 Hours of Preoperative Fasting in Breast-feeding Infants
Acronym: BMRCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University Hospital (Other)
Responsible Party: Principal Investigator, Peter Frykholm, Assoc. Prof., Uppsala University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMRCT PILOT
Record Dates: First submitted 2022-09-02; First posted 2022-10-10 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Perioperative Complication
Keywords: Preoperative fasting; Anaesthesia; Children; breast-feeding
MeSH Terms: conditions — Breast Feeding | interventions — Milk, Human

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled pilot study
Who Masked: Investigator, Outcomes Assessor
Masking Description: Computerized randomization,
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3h Group (Experimental): the patient's parents are instructed to stop feeding 3 hours for scheduled anesthesia. (3 hours of preoperative fasting for breast milk)
  Interventions: Other: 3 hours of preoperative fasting for breast milk
- 4h Group (Active Comparator): the patient's parents are instructed to stop feeding 4 hours for scheduled anesthesia (4 hours of preoperative fasting for breast milk)
  Interventions: Other: 4 hours of preoperative fasting for breast milk

INTERVENTIONS:
Other: 3 hours of preoperative fasting for breast milk — 3 hours of preoperative fasting for breast milk
  Arms: 3h Group
Other: 4 hours of preoperative fasting for breast milk — 4 hours of preoperative fasting for breast milk
  Arms: 4h Group

SUMMARY:
In the new guideline from ESAIC breast-feeding should be encouraged until 3 hours before anesthesia. This recommendation was based mainly on gastric emptying studies in neonates with small sample sizes and single center experience.To address the lack of high quality evidence for this recommendation, the ESAIC task force for preoperative fasting plans perform a multicenter RCT omparing 4 vs 3 hours of preoperative fasting for breast milk.

The aim of the present pilot-study is to provide data for sample size calculation and feasibility for the multicenter trial.

DETAILED DESCRIPTION:
Since the publication of several studies indicating that many children are subjected to unnecessarily long fasting waiting for surgery, there is great interest within the pediatric anesthesia community to understand gastric emptying to be able to revise existing guidelines. The new recommendation from ESAIC is that breast-feeding should be encouraged until 3 hours before anesthesia. This recommendation was based mainly on gastric emptying studies in neonates with small sample sizes and single center experience.To address the lack of high quality evidence for this recommendation, the task force plans to perform a multicenter RCT comparing 4 vs 3 hours of preoperative fasting for breast milk.

Twenty infants scheduled for elective surgery or procedures requiring general anesthesia or sedation will be recruited for this randomized controlled pilot study.

Based on the randomization, they are then asked to breast-feed (or bottle-feed with breast-milk) the child at 4 or 3 hours before the scheduled anesthesia induction.

On arrival to the operating room, the gastric ultrasound examination will be performed for analysis of the gastric antrum CSA. After i.v. or inhalational anesthesia, an oro-gastric catheter will be inserted and any residual gastric contents are aspirated when rotating the infant from supine to semi-prone right and left positions. The volume and color of the aspirate will be recorded.

The aim of the present pilot-study is to provide data for sample size calculation and feasibility for the multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

- Breast-feeding infanta scheduled for elective procedure requiring general anesthesia

Exclusion Criteria:

* infant that does not breast-feed or is bottle-fed breast-milk
* Moderate to severe gastrointestinal motility disorder.
* Emergency surgery.
* Age > 24 months or age < 37 gestational weeks
* parents incapable of understanding the consent information due to language barrier

Ages: 0 Years to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
CSA | From arrival in the operating room until induction of anesthesia
  Gastric antrum CSA (The antral cross-sectional area)

SECONDARY OUTCOMES:
Aspirated volume | intraoperative
  Aspirated volume

CONTACTS AND LOCATIONS:
Overall Officials: Peter Frykholm, MD, PhD, Principal Investigator — Uppsala University Hospital
Locations (1):
- Uppsala University Hospital, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pre-operative fasting in children: A guideline from the European Society of Anaesthesiology and Intensive Care — https://pubmed.ncbi.nlm.nih.gov/34857683/
- See also: Gastric content assessed with gastric ultrasound in paediatric patients prescribed a light breakfast prior to general anaesthesia: A prospective observational study — https://pubmed.ncbi.nlm.nih.gov/31608517/
- See also: Ultrasound assessment of gastric emptying time after intake of clear fluids in children scheduled for general anesthesia-A prospective observational study — https://pubmed.ncbi.nlm.nih.gov/32997821/